CLINICAL TRIAL: NCT03678220
Title: Clinical Translation of Augmented Reality Visualization for Laparoscopic Surgery
Brief Title: Assessment of Augmented Reality in Minimally Invasive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IGI Technologies, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LAPAR01; 2R42CA192504 (NIH)
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-09

CONDITIONS: Laparoscopic Hepatectomy; Laparoscopic Liver Thermal Ablation
Keywords: Laparoscopic Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients using LapAR system (Experimental)
  Interventions: Device: LapAR

INTERVENTIONS:
Device: LapAR — LapAR system will be used for guidance during laparoscopic hepatectomy and laparoscopic liver thermal ablation

SUMMARY:
The objective of this study is to test the technical feasibility of LapAR visualization system for guiding laparoscopic surgeries and to gather clinical feedback on the use of this tool.

DETAILED DESCRIPTION:
Surgeons use real-time video generated by a laparoscope to visualize the operative field when performing laparoscopic procedures. An inability to see beneath organ surfaces is a limitation of the current visualization technology. Surgeons additionally use laparoscopic ultrasound to see beneath organ surfaces, but also need to mentally correlate the ultrasound image with the video of the operative field. This process is difficult, subjective, and variable with expertise, and discourages the use of ultrasound.

The investigators have developed a method to combine live laparoscopic video and laparoscopic ultrasound images to present fused multimodality images on a single display, eliminating the need for mental image correlation. Specifically, the image fusion method, called laparoscopic augmented reality (LapAR), augments the laparoscopic video with ultrasound data when required by surgeons. This study is designed to test this minimal-risk capability in patients referred for relevant laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is referred for either laparoscopic partial hepatectomy for tumor removal or laparoscopic ablation of liver cancer;
2. Patient must be at least 18 years old;
3. Patient provides written consent;
4. Patient is considered a suitable candidate based on tumor location for using the AR system.

Exclusion Criteria:

Patients with pacemaker or any other ICD(intra-cardiac device) which may interfere with electromagnetic tracking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Surgeon interview regarding usability | post surgery, an expected average of 5 minutes
  The ease of use of the LapAR system will be evaluated by the surgeon
Procedure time | during surgery
  Time of using the LapAR system for laparoscopic hepatectomy and laparoscopic thermal ablation
Measurement of margin | post surgery
  Obtain from Pathology department or follow-up imaging

SECONDARY OUTCOMES:
System set-up time | before surgery, an expected average of 15 min

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States